CLINICAL TRIAL: NCT07185139
Title: Exploratory Clinical Trial of MSCohi-O Lenses for Ocular Involvement in Sjögren's Syndrome
Brief Title: MSCohi-O Lenses for Ocular Involvement in Sjögren's Syndrome
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLKR-MSCohi-O-501
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sjögren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCohi-O Lenses Group (Experimental): Each subject will wear MSCohi-O Lenses for 12 hours a day, totally 14-day wearings.
  Interventions: Drug: MSCohi-O Lenses

INTERVENTIONS:
Drug: MSCohi-O Lenses — Each subject will wear MSCohi-O Lenses for 12 hours a day, totally 14 wearings.
  Other Names: MSCohi-O

SUMMARY:
This study is aSingle-center, multiple-dosing, prospective, nonrandom, single-arm trial.

DETAILED DESCRIPTION:
This study is aSingle-center, multiple-dosing, prospective, nonrandom, single-arm trial. To evaluate the clinical safety and efficacy of MSCohi-O Lenses in patients with ocular involvement of Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old, including the boundary value, no gender restriction;
* Subjects meeting the 2016 ACR/EULAR classification criteria for Sjögren's syndrome, and also meet the diagnostic criteria for ocular involvement.
* Ocular signs and symptoms unresponsive to at least 3 months of conventional therapy, including artificial tears and topical or systemic corticosteroids.
* Extra-ocular manifestations of Sjögren's syndrome clinically stable.
* Subjects and their partners agree to use effective non-pharmacological contraception from screening through 6 months after the last dose and have no plans for conception during this period.
* Willing to participate in the study, understand and sign the informed consent form (ICF).

Exclusion Criteria:

* Known allergy to any component of the investigational drug.
* Active ocular infection.
* Presence of other significant ocular disease or trauma diagnosed prior to enrollment, including but not limited to glaucoma, uveitis, retinopathy, chemical injury, or thermal burns.
* History of any ocular surgery within the preceding 6 months, including cataract surgery.
* Participation in another interventional clinical study.
* Use of any ophthalmic medication that may interfere with the study outcomes, such as other stem-cell-derived products.
* Having serious underlying diseases of the heart, brain vessels, liver, kidneys, and hematopoietic system.
* Pregnant or lactating women; women of childbearing potential must employ an effective contraceptive method (e.g., intrauterine device, oral contraceptive, or condom) during the study and for at least 3 months after the final dose of study drug.
* Subjects deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | from subjects receiving administration to Day 29 post-administration
  Incidence and severity of adverse events from subjects receiving administration to Day 29 post-administration.

SECONDARY OUTCOMES:
corneal fluorescein staining | from baseline to Day 8, Day 15 and Day 29 post-administration
  Changes in corneal fluorescein staining scores from baseline to Day 8, Day 15 and Day 29 post-administration.
Tear film break-up time | from baseline on Day 8, Day 15 and Day 29 post-administration
  Changes in Tear film break-up time from baseline on Day 8, Day 15 and Day 29 post-administration.
ocular surface disease index scores | from baseline on Day 8, Day 15 and Day 29 post-administration
  Changes in ocular surface disease index scores from baseline on Day 8, Day 15 and Day 29 post-administration
Schirmer's test | from baseline on Day 8, Day 15 and Day 29 post-administration
  Changes in Schirmer's test from baseline on Day 8, Day 15 and Day 29 post-administration.

IPD SHARING:
Plan to Share IPD: No